CLINICAL TRIAL: NCT02349594
Title: Modulation of Immune Function by Parenteral Fish Oil in Patients With Crohn's Disease and High Inherent Tumor Necrosis Factor-alpha Production: a Randomized, Single Blinded, Cross-over Study
Brief Title: Immune Modulation by Parenteral Fish Oil in Patients With Crohn's Disease
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Treatment
Other Study IDs: GW/MB/42964; 2013-001212-30 (EudraCT Number)
Record Dates: First submitted 2015-01-16; First posted 2015-01-29 (Estimated); Last update posted 2015-11-10 (Estimated); Status verified 2015-11

CONDITIONS: Crohn Disease
MeSH Terms: conditions — Crohn Disease | interventions — Fish Oils; Soybean Oil

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- treatment order A (Active Comparator): Participants in this arm first receive 'Omegaven 10%' and after crossing over the 'Intralipid 20%'
  Interventions: Drug: Omegaven 10%; Drug: Intralipid 20%
- treament order B (Active Comparator): Participants in this arm first receive 'Intralipid 20%' and after crossing over the 'Omegaven 10%'
  Interventions: Drug: Omegaven 10%; Drug: Intralipid 20%

INTERVENTIONS:
Drug: Omegaven 10% — intravenous administration 10% (w/v) fish oil emulsion (Omegaven) for 1 hour on three consecutive days at a dose of 0.2 g/kg bodyweight/hr.
  Other Names: fish oil; N-3 polyunsaturated fatty acids atty acids
Drug: Intralipid 20% — intravenous administration of 20% (w/v) lipid-control (Intralipid®), for 1 hour on three consecutive days at a dose of 0.2 g/kg bodyweight/hr.
  Other Names: soybean oil; N-6 polyunsaturated fatty acids atty acids

SUMMARY:
To evaluate the effects of infusion of a Fish oil-based lipid emulsion on TNF-α production and other relevant immune functions. A soybean oil emulsion, rich in the omega-6 polyunsaturated fatty acid linoleic acid, will serve as control.

DETAILED DESCRIPTION:
Rationale: Fish oil (FO), rich in omega-3 polyunsaturated fatty acids, exerts a range of anti-inflammatory actions that render it a potential therapeutic agent to treat Crohn's disease, a chronic inflammatory disease that primarily affects the bowel. Recent evidence suggests that a lack of effect in previous studies might be due to the fact that genetic background was not taken into account. For instance, a study in healthy subjects showed that production of the pro-inflammatory cytokine Tumor Necrosis Factor-alpha (TNF-α) following FO supplementation decreased in individuals within the highest tertile of pre-supplementational TNF-α production, remained unaltered in the middle tertile, and increased in the lowest tertile of pre-supplementational TNF-α production. TNF-α plays a pivotal role in the pathogenesis of Crohn's disease, hence the treatment with anti-TNF-α agents. Based on these notions, and because FO supplementation via the enteral route is strongly dose limited due to fat-induced side effects such as diarrhea, we hypothesize that parenteral FO supplementation might be beneficial in those patients with Crohn's disease with a high inherent TNF-α production.

Study design: Single center, randomized, single blinded, lipid-controlled, cross-over pilot trial.

Study population: Adult patients with Crohn's disease with previous bowel surgery, currently in remission (without the need for immunosuppressive drugs) and with a high inherent TNF-α production.

Intervention: First, patients with a high inherent TNF-α will be identified by assessment of TNF-α production in a group 100 patients who meet in- and exclusion criteria. Patients within the highest tertile will be classified as high producers. Next, 5 patients within the highest tertile will be randomized to receive intravenous administration of 20% (w/v) lipid-control (Intralipid®), and, after crossing over, 10% (w/v) fish oil emulsion (Omegaven®), or vice-versa for 1 hour on three consecutive days at a dose of 0.2 g/kg bodyweight /hr. Study parameters will be assessed in blood drawn prior to the first infusion (T=0) and 1 (T=4) and 8 days (T=11) after the third infusion. Between the two treatment arms, there will be a wash-out interval of at least 2-3 weeks.

Main study parameters/endpoints: Early (T=day 4) and late (T=day 11) effects of infusions on TNF-α production by whole blood cultures. Secondary outcomes: effect on leukocyte counts, leukocyte functions and on (anti-)oxidant status, the occurrence of oxidative damage and analysis of specific Single Nucleotide Polymorphisms (SNPs) related to TNF-α production.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients with Crohn's disease with previous bowel surgery, currently in remission (without the need for immunosuppressive drugs) and with a high inherent TNF-α production.

Exclusion Criteria:

* Patients with other active inflammatory / immune mediated underlying diseases
* Smoking > 5 cigarettes a day
* Diet with >2 portions of fatty fish (tuna, salmon, mackerel, herring, and trout) a week
* History of metabolic disorder (especially diabetes or lipid disorders)
* Crohn's disease activity, including the presence of active fistulas
* On need for medical (other than 5-aminosalicylic acid preparations) or surgical treatment for Crohn's disease activity
* Use of non-steroidal anti-inflammatory drugs or aspirin
* C-reactive protein levels of >10 mg/l
* History of venous or arterial thrombosis
* Active malignancy
* Presence of severe pulmonary, cardiovascular, renal, liver, coagulation or hematological disease
* Pregnancy or lactation
* Age <18 yrs
* Allergy for one of the following components: fish, chicken, eggs or soy beans

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2014-01; Primary Completion 2015-05 (Actual); Study Completion 2015-09 (Actual)

PRIMARY OUTCOMES:
Change of TNF-α production in pg/ml | day 0 and day 4
  whole blood cultures are stimulated with 1 ng/ml lipopolysaccharide for 4 hours. TNF-alpha levels are measured in the supernatant with an enzyme-linked immunosorbent assay. Differences are compared by paired t-test or wilcoxon signed rank test.

SECONDARY OUTCOMES:
short term change in leukocyte functions | day 0 and day 4
  Change in expression of cell surface markers on neutrophils and monocytes (CD11, CD66, CD62 and CD63) by immune fluorescent staining and subsequent flowcytometric analysis. Between day 0 and day 4 patients receive on intralipid or omegaven 3 consecutive days. Differences are compared by paired t-test or wilcoxon signed rank test
long term change in leukocyte functions | day 0 and day 11
  Change in expression of cell surface markers on neutrophils and monocytes (CD11, CD66, CD62 and CD63) by immune fluorescent staining and subsequent flowcytometric analysis. Differences are compared by paired t-test or wilcoxon signed rank test.
change in Oxygen radical production by neutrophils | day 0 and day 4
  Differences are compared by paired t-test or wilcoxon signed rank test
change in Oxygen radical production by neutrophils | day 0 and day 11
  Differences are compared by paired t-test or wilcoxon signed rank test.
short term effects on in cytokine production | day 0 and day 4
  whole blood cultures are stimulated with 1 ng/ml lipopolysaccharide for 24 hours. Interleukin (IL)-1B, Il-6 and IL-10 levels are measured in the supernatant with an enzyme-linked immunosorbent assay. Differences are compared by paired t-test or wilcoxon signed rank test.
Long term effects on in cytokine production | day 0 and day 11
  whole blood cultures are stimulated with 1 ng/ml lipopolysaccharide for 24 hours. Il-1B, Il-6 and IL-10 levels (pg/ml ) are measured in the supernatant with an enzyme-linked immunosorbent assay . Differences are compared by paired t-test or wilcoxon signed rank test.
Composition of phospholipids in the cell membrane | day 0, day4 and day 11
  to evaluate fatty acid incorporationDifferences are compared by paired t-test or wilcoxon signed rank test.
Change of TNF-α production in pg/ml | day 0 and day 11
  whole blood cultures are stimulated with 1 ng/ml lipopolysaccharide for 4 hours. TNF-alpha levels are measured in the supernatant with an enzyme-linked immunosorbent assay. Differences are compared by paired t-test or wilcoxon signed rank test.
(anti-) Oxidant status and oxidative damage | day 0 and day 4
  Oxidative stress will be measured by both lipid and protein peroxidation and antioxidant capacity. Differences are compared by paired t-test or wilcoxon signed rank test.
(anti-) Oxidant status and oxidative damage | day 0 and day 11
  Oxidative stress will be measured by both lipid and protein peroxidation and antioxidant capacity. Differences are compared by paired t-test or wilcoxon signed rank test.

CONTACTS AND LOCATIONS:
Overall Officials: G. Wanten, MD, PhD, Study Director — Radboud University Nijmegen Medical Center; F. Hoentjen, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center; D de Jong, MD, PhD, Principal Investigator — Radboud University Nijmegen Medical Center; P. Calder, MD, PhD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (1):
- Radboud University Medical Center, Nijmegen, Netherlands